CLINICAL TRIAL: NCT00487994
Title: A Double-Blind, Randomized, Parallel Group Study to Evaluate the Safety, Tolerability and Efficacy of Lapaquistat Acetate Alone or Coadministered With Atorvastatin in Subjects With Primary Dyslipidemia
Brief Title: Safety and Efficacy of Lapaquistat Acetate Taken Alone and With Atorvastatin in Subjects With Primary Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-475-002; 2004-000775-34 (EudraCT Number); U1111-1122-7619 (Registry Identifier: WHO)
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Dyslipidemia
Keywords: Hypercholesterolemia; Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lapaquistat Acetate 100 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Lapaquistat Acetate 100 mg QD + Atorvastatin 10 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate and atorvastatin
- Atorvastatin 10 mg QD (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate — Lapaquistat acetate 100 mg, tablets, orally, once daily and Atorvastatin placebo-matching capsules, orally, once daily for up to 96 weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD
Drug: Lapaquistat acetate and atorvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and Atorvastatin 10 mg, capsules, orally, once daily for up to 96 weeks.
  Other Names: TAK-475; Lipitor
  Arms: Lapaquistat Acetate 100 mg QD + Atorvastatin 10 mg QD
Drug: Atorvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and Atorvastatin 10 mg, capsules, orally, once daily for up to 96 weeks.
  Other Names: Lipitor
  Arms: Atorvastatin 10 mg QD

SUMMARY:
The purpose of this study is to evaluate the overall safety of Lapaquistat Acetate, once daily (QD), by itself or in combination with atorvastatin in subjects with primary dyslipidemia.

DETAILED DESCRIPTION:
According to the World Health Organization, CHD is now the leading cause of death worldwide. In 2001, CHD caused 7.2 million deaths and estimates for 2020 indicate that annual CHD deaths will increase to 11.1 million. These statistics suggest that improved options are needed to treat hypercholesterolemia and dyslipidemia.

The balance among cholesterol synthesis, dietary intake, and degradation is normally adequate to maintain healthy cholesterol plasma levels. However, in patients with hypercholesterolemia, elevated low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls. Consequently, in this population it has been established that lowering low-density lipoprotein cholesterol plasma concentrations effectively reduces cardiovascular morbidity and mortality. The National Cholesterol Education Program Adult Treatment Panel III has therefore identified control of low-density lipoprotein cholesterol as essential in the prevention and management of CHD. Additional lipid risk factors designated by National Cholesterol Education Program Adult Treatment Panel III include elevated triglycerides, elevated non-high-density lipoprotein cholesterol (atherogenic lipoproteins), and low levels of high-density lipoprotein cholesterol. Lipoproteins rich in triglycerides, such as very-low-density lipoprotein cholesterol, appear to contribute to atherosclerosis, whereas the apparent protective effect of high-density lipoprotein cholesterol, which is likely related to high-density lipoprotein cholesterol-facilitated transport of cholesterol away from atherosclerotic deposits, may be limited at low high-density lipoprotein cholesterol concentrations.

Initial dietary and lifestyle measures taken to control dyslipidemia are often inadequate, and most patients require pharmacologic intervention. Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (statins) are the first-line monotherapies most often prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, with statin monotherapy, many patients fail to reach National Cholesterol Education Program Adult Treatment Panel III recommended levels of low-density lipoprotein cholesterol reduction. As a result, the statin dosage must be increased or an additional treatment added to achieve treatment goals. Increasing the statin dosage may result in decreased tolerability and potential safety concerns, contributing to the high discontinuation rates of statins and their prescription at low and often ineffective doses. Further, although the effectiveness of increasing the dose varies among the statins, in general, doubling of the dose above the minimum effective dose has been found to decrease serum low-density lipoprotein cholesterol by only an additional 6 percent.

TGRD is developing an orally active squalene synthase inhibitor, TAK-475 (lapaquistat acetate) for the treatment of dyslipidemia. Lapaquistat acetate inhibits the biosynthesis of cholesterol by inhibiting the enzyme squalene synthase, which catalyzes the conversion of farnesyl diphosphate to squalene-a precursor in the final steps of cholesterol production.

Study Participation is anticipated to be up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmatory central laboratory result with low density lipoprotein cholesterol greater than or equal to 3.37 mmol/L and less than 5.69 mmol/L, and triglyceride less than 4.52 mmol/L.
* Females of child-bearing age must have undergone surgical sterilization, hysterectomy, tubal ligation, or bilateral oophorectomy; other female subjects must have been postmenopausal.
* Must be in good physical and mental health as determined by a physician on the basis of medical history, physical examination, and laboratory results.
* Has a fasting low density lipoprotein cholesterol level greater than or equal to 3.37 mmol/L and less than 4.92 mmol/L, and a triglyceride value less than 4.52 mmol/L.

Exclusion Criteria:

* Coronary Heart Disease or Coronary Heart Disease-risk factors comprised of:

  * Diabetes mellitus type 1 or 2.
  * History or presence of myocardial infarction, angina pectoris, unstable angina, coronary angioplasty, coronary or peripheral arterial surgery (bypass graft), aortic aneurysm, transient ischemic attacks, or cerebrovascular accident.
* A body mass index less than 15 or greater than 35.
* A history or presence of:

  * Drug abuse or a history of alcohol abuse within the 2 years previous to screening.
  * Uncontrolled hypertension despite medical treatment
  * Thyroid disease, particularly hyperthyroidism or subjects whose thyroid replacement therapy was initiated within the previous 3 months.
  * Human immunodeficiency virus-positive status, or hepatitis B or C infection.
  * Malignancy, except subjects whose malignancy had been diagnosed as stage I basal or squamous cell carcinoma.
  * Heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia.
  * Fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain and/or discontinuation of statins due to myalgia.
  * Trauma to the eye or eye irradiation; glaucoma; iritis; uveitis; prior intraocular surgery, laser surgery to the iris, retinal photocoagulation, or laser trabeculoplasty; corneal opacification or other medial opacities; or had undergone LASIK refractive surgery within 6 months prior to screening.
  * A clinically significant food allergy that would prevent adherence to the specialized diet.
* Any other serious disease or condition that might have affected life expectancy or made it difficult to successfully manage and monitor the subject according to the protocol.
* Has a known hypersensitivity or history of adverse reaction to atorvastatin or to lapaquistat acetate.
* Is taking part in another investigational study or had been participating in an investigational study within the 30 days prior to Screening Visit 1.
* Has an alanine aminotransferase or aspartate aminotransferase level greater than 2 times the upper limit of normal, active liver disease, jaundice, serum creatinine greater than 135 μmol/L (1.5 mg/dL), or creatine kinase greater than 3 times the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2130 (Actual)
Dates: Start 2004-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Lens Opacity Classification System findings | Weeks 24, 48, 72, and 96 or Final Visit
Best corrected visual acuity | Weeks 24, 48, 72, and 96 or Final Visit
Adverse Events | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96 or Final Visit
Clinical Laboratory Tests | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96 or Final Visit
Vital signs (blood pressure and pulse rate) and weight | Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96 or Final Visit
12-lead Electrocardiogram | Weeks 48 and 96 or Final Visit
Physical Examination | Weeks 48 and 96 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Low Density Lipoprotein cholesterol | Week 96 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 96 or Final Visit
Change from Baseline in Total Cholesterol | Week 96 or Final Visit
Change from Baseline in Triglycerides | Week 96 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 96 or Final Visit
Change from Baseline in Apolipoprotein A1 | Week 96 or Final Visit
Change from Baseline in Apolipoprotein B | Week 96 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (128):
- United States (61):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Northport, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Sierra Vista, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Rancho Cucamonga, California
  - Santa Rosa, California
  - Golden, Colorado
  - Coral Gables, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Sarasota, Florida
  - West Palm Beach, Florida
  - Dunwoody, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Waterloo, Iowa
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Flint, Michigan
  - Edina, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Ship Bottom, New Jersey
  - Rochester, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Tipton, Pennsylvania
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Cordova, Tennessee
  - Morristown, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Texarkana, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
- Argentina (8):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Morón
  - Pilar
  - Rosario
  - Salta
  - Santa Fe
- Santiago, Chile
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Tartu, Estonia
- Germany (8):
  - Berlin
  - Freiburg im Breisgau
  - Görlitz
  - Hamburg
  - Mannheim
  - Mönchengladbach
  - Munich
  - Schwerin
- Hungary (7):
  - Budapest
  - Debrecen
  - Esztergom
  - Győr
  - Gyula
  - Kecskemét
  - Warszawa
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Vilnius
  - Vilnius-21
- Mexico (6):
  - Distrito Federal
  - Guadalajara
  - Jalisco
  - Mexico City
  - San Luis Potosí City
  - Zapopan
- Netherlands (5):
  - Es Velp
  - Groningen
  - Leiden
  - Rotterdam
  - Zoetermeer
- Lima, Peru
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Gorzów Wielkopolski
  - Grudziądz
  - Płońsk
  - Torun
  - Wroclaw
  - Włocławek
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- Slovakia (3):
  - Komárno
  - Košice
  - Levice
- South Africa (4):
  - Cape Town
  - Johannesburg
  - Parow
  - Western Cape
- United Kingdom (4):
  - Truro, Cornwall
  - Blackpool, Lancashire
  - Bolton, Lancashire
  - Guildford, Surrey

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985